CLINICAL TRIAL: NCT05388539
Title: TBS Treatment for Treatment-Resistant Depression: a Randomized, Sham-Controlled Trial
Brief Title: TBS Treatment for Treatment-Resistant Depression
Acronym: TTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Andre R Brunoni, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 52384921.6.0000.0068
Record Dates: First submitted 2022-05-13; First posted 2022-05-24 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder; Unipolar Depression
Keywords: Unipolar Depression; Major Depressive Disorder; Transcranial Magnetic Stimulation; Neuromodulation; Theta Burst Stimulation; Accelerated Theta Burst Stimulation; Intermittent Theta Burst Stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group - protocol of Theta Burst Stimulation (Active Comparator): 3 sessions of theta burst stimulation, 1200 pulses per session of 6 minutes duration, 30-minute interval between sessions. Stimulation directed to the left dorsolateral pre-frontal cortex. The protocol will be applied for 15 days, totalizing 45 sessions of stimulation.
  Interventions: Procedure: Theta Burst Stimulation
- Placebo Group - Sham Stimulation (Placebo Comparator): The placebo will consist of a sham stimulation activity. A noise generator, which makes the same noise as active stimulation, and a surface electrode placed over the patient's eyebrow, mimicking the tactile sensory effects of TBS.
  Interventions: Procedure: Sham Stimulation

INTERVENTIONS:
Procedure: Theta Burst Stimulation — 3 TBS sessions per day, with an offer of 1200 pulses per session and a 30-minute interval between sessions. This protocol will be applied to patients for 15 days, totaling 45 stimulation sessions. The stimulations will be directed to the left dorsolateral prefrontal cortex (F3 obtained by the Beam method) and will be performed in a Magventure MagPro R30 device.The stimulation will be delivered at 100% of the motor threshold and will last for 6 minutes.
  Other Names: Transcranial Magnetic Stimulation; Magventure - MagPro R30
  Arms: Active Group - protocol of Theta Burst Stimulation
Procedure: Sham Stimulation — The placebo will consist of a sham stimulation activity. A noise generator, which makes the same noise as active stimulation, and a surface electrode placed over the patient's eyebrow, mimicking the tactile sensory effects of TBS. It will also occur three times a day, with a duration of 6 minutes. The interval time between procedures will be of 30 minutes. It will take place for the same 15 weekdays, totalizing 45 sham stimulations.
  Other Names: Placebo/Sham Stimulation
  Arms: Placebo Group - Sham Stimulation

SUMMARY:
Depression is a highly disabling disease that is prevalent throughout the world. The treatments proposed and studied to date have shown to be partially effective in treating this condition. Neuromodulation strategies have been used as an alternative, especially for refractory and challenging cases. In this context, studies investigating the effectiveness of transcranial magnetic stimulation, including the theta burst stimulation (TBS) modality, have been increasing in number. However, there is still a lack of information seeking to explore the maximum effectiveness in the TBS modality. Therefore, the investigators developed a new stimulation protocol consisting of 3 TBS sessions per day, with an offer of 1200 pulses per session and a 30-minute interval between sessions. The protocol will be performed for 15 days, totalizing 45 stimulation sessions. The stimulations will be directed to the left dorsolateral prefrontal cortex (F3) and will be performed in a Magventure MagPro R30 device. The investigators will select 100 patients with unipolar major depression, following previously established inclusion and exclusion criteria, and will apply the protocol randomly, dividing the patients into an active and placebo group. The research team hypothesized that the active group patients will have greater improvement in symptoms of depression assessed by the 17-item hamilton depression scale over patients of the placebo group. In addition, other scales will be used for secondary outcomes. The researchers also hypothesized that there will be no difference between patients placed in the active or placebo groups in terms of side effects.

DETAILED DESCRIPTION:
Depression is a highly disabling disease that is prevalent throughout the world. The treatments proposed and studied to date have shown to be partially effective in treating this condition. Neuromodulation strategies have been used as an alternative, especially for refractory and challenging cases. In this context, studies investigating the effectiveness of transcranial magnetic stimulation, including the theta burst stimulation (TBS) modality, have been increasing in number. However, there is still a lack of information seeking to explore the maximum effectiveness in the TBS modality. Therefore, the investigators developed a stimulation protocol consisting of 3 TBS sessions per day, with an offer of 1200 pulses per session and a 30-minute interval between sessions. This protocol will be applied to patients for 15 days, totaling 45 stimulation sessions. The stimulations will be directed to the left dorsolateral prefrontal cortex (F3 obtained by the Beam method) and will be performed in a Magventure MagPro R30 device.

The stimulation will be delivered at 100% of the motor threshold and will last for 6 minutes. The placebo will consist of a noise generator, which makes the same noise as active stimulation, and a surface electrode placed over the patient's eyebrow, mimicking the tactile sensory effects of TBS. The researchers will select 100 patients with unipolar major depression, following previously established inclusion and exclusion criteria, and the protocol will be applied randomly, dividing the patients into an active and placebo group. Inclusion criteria are: patients with a diagnosis of unipolar major depression confirmed by the Mini International Neuropsychiatric Interview (MINI), between 18 and 59 years of age, with a Hamilton score equal to or greater than 17. In addition, patients must have undergone at least 1 first-line treatment for depression and a maximum of 3 previous unsuccessful treatments. Exclusion criteria are: other mental disorders (bipolar affective disorder, obsessive-compulsive disorder, attention deficit hyperactivity disorder, personality disorders, substance use disorder, psychotic disorders), history of suicide attempts or severe suicidal ideation in the last 6 months. In addition, patients who have a history of epilepsy, decompensated medical conditions, metallic implants in the skull or previous experience with transcranial magnetic stimulation will be excluded.

The investigators hypothesized greater improvement in the symptoms of depression in patients of the active group compared with the placebo group, assessed by the 17-item hamilton depression scale. In addition, other scales for secondary outcomes wil be used, such as the Montgomery-Asberg Depression Scale. The research team also hypothesized that there will be no difference between patients in the different groups in terms of side effects. In the patient selection process, individuals will be evaluated and submitted to questionnaires in consultations by video call with a medical doctor of the research team. During the study, patients will be evaluated weekly and in person, by professionals who are not part of the stimulation application group. The service's waiting room will be organized in a certain way, so that patients do not meet or communicate during the study. After the end of the stimulations, the patients will be followed up for another 2 weeks in order to evaluate the support of the response obtained during the investigation. All data will be stored in a secure database with an external hard drive. All ethical considerations will be discussed with patients and followed during the study. The project has already been approved by the ethics committee of the Hospital of Clinics of the University of Sao Paulo. A pilot study will be conducted to assess the feasibility of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are: patients with a diagnosis of unipolar major depression confirmed by the MINI interview, between 18 and 59 years of age, with a Hamilton score equal to or greater than 17. In addition, patients must have undergone at least 1 first-line treatment for depression and a maximum of 3 previous unsuccessful treatments.

Exclusion Criteria:

* Exclusion criteria are: other mental disorders (bipolar affective disorder, obsessive-compulsive disorder, attention deficit hyperactivity disorder, personality disorders, substance use disorder, psychotic disorders), history of suicide attempts or severe suicidal ideation in the last 6 months. In addition, patients who have a history of epilepsy, decompensated medical conditions, metallic implants in the skull or previous experience with transcranial magnetic stimulation will be excluded.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (17 Items) | 5 weeks
  Scale to assess depressive symptoms - The minimum scale score is 0 and the maximum scale score is 50 points. The standardized scores are: 7 to 17 points - mild depression; 18 to 25 points - moderate depression and 26 or more points - severe depression. Higher scores mean worse clinical condition or outcome.

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale | 5 weeks
  Scale to assess depressive symptoms The minimum scale score is 0 and the maximum scale score is 60 points. The standardized scores are: 7 to 19 points - mild depression; 20 to 34 points - moderate depression and 35 or more points - severe depression. Higher scores mean worse clinical condition or outcome.
Collateral Effects Rating Scale | 5 weeks
  Scale to assess side effects of the procedure - not a numeric scale. It consist of a scale to assess the severity of side effects between: absent, mild, moderate and severe. In addition, the investigators seek to correlate the possible side effect with the procedure in the face of the following alternatives: remotely related, possibly related, probably related, certainly related. For this, the patient's own report, will be taken into account.

CONTACTS AND LOCATIONS:
Overall Officials: Andre R Brunoni, MD, PhD, Study Director — University of Sao Paulo
Locations (1):
- Institute of Psychiatry - University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Participant data can only be accessed by study members. Such data will be stored in a database with an external hard drive (HD). The only way to access this database is to be affiliated with the institution where the study will be conducted and to request authorization from the study director, who coordinates access for the other researchers.
  During the study, each participant will be evaluated by a single professional and this professional from the research group will be the only one with conditions to add or change clinical data according to evaluation.
  After data analysis and the end of the research, supplementary materials containing a database preserving the anonymity of the participants will be made available.

REFERENCES:
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Carvalho AF, Sharma MS, Brunoni AR, Vieta E, Fava GA. The Safety, Tolerability and Risks Associated with the Use of Newer Generation Antidepressant Drugs: A Critical Review of the Literature. Psychother Psychosom. 2016;85(5):270-88. doi: 10.1159/000447034. Epub 2016 Aug 11. PMID 27508501
- [Background] Meyer JP, Swetter SK, Kellner CH. Electroconvulsive Therapy in Geriatric Psychiatry: A Selective Review. Psychiatr Clin North Am. 2018 Mar;41(1):79-93. doi: 10.1016/j.psc.2017.10.007. Epub 2017 Dec 13. PMID 29412850
- [Background] Wischnewski M, Schutter DJ. Efficacy and Time Course of Theta Burst Stimulation in Healthy Humans. Brain Stimul. 2015 Jul-Aug;8(4):685-92. doi: 10.1016/j.brs.2015.03.004. Epub 2015 Mar 26. PMID 26014214
- [Background] McClintock SM, Reti IM, Carpenter LL, McDonald WM, Dubin M, Taylor SF, Cook IA, O'Reardon J, Husain MM, Wall C, Krystal AD, Sampson SM, Morales O, Nelson BG, Latoussakis V, George MS, Lisanby SH; National Network of Depression Centers rTMS Task Group; American Psychiatric Association Council on Research Task Force on Novel Biomarkers and Treatments. Consensus Recommendations for the Clinical Application of Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Depression. J Clin Psychiatry. 2018 Jan/Feb;79(1):16cs10905. doi: 10.4088/JCP.16cs10905. PMID 28541649
- [Background] Berlim MT, McGirr A, Rodrigues Dos Santos N, Tremblay S, Martins R. Efficacy of theta burst stimulation (TBS) for major depression: An exploratory meta-analysis of randomized and sham-controlled trials. J Psychiatr Res. 2017 Jul;90:102-109. doi: 10.1016/j.jpsychires.2017.02.015. Epub 2017 Feb 21. PMID 28254709
- [Background] Brunoni AR, Chaimani A, Moffa AH, Razza LB, Gattaz WF, Daskalakis ZJ, Carvalho AF. Repetitive Transcranial Magnetic Stimulation for the Acute Treatment of Major Depressive Episodes: A Systematic Review With Network Meta-analysis. JAMA Psychiatry. 2017 Feb 1;74(2):143-152. doi: 10.1001/jamapsychiatry.2016.3644. PMID 28030740
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, Nejad R, Pankow H, Choi E, Aaron H, Espil FM, Pannu J, Xiao X, Duvio D, Solvason HB, Hawkins J, Guerra A, Jo B, Raj KS, Phillips AL, Barmak F, Bishop JH, Coetzee JP, DeBattista C, Keller J, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020 Aug 1;177(8):716-726. doi: 10.1176/appi.ajp.2019.19070720. Epub 2020 Apr 7. PMID 32252538
- [Background] Brunoni AR, Moffa AH, Sampaio-Junior B, Borrione L, Moreno ML, Fernandes RA, Veronezi BP, Nogueira BS, Aparicio LVM, Razza LB, Chamorro R, Tort LC, Fraguas R, Lotufo PA, Gattaz WF, Fregni F, Bensenor IM; ELECT-TDCS Investigators. Trial of Electrical Direct-Current Therapy versus Escitalopram for Depression. N Engl J Med. 2017 Jun 29;376(26):2523-2533. doi: 10.1056/NEJMoa1612999. PMID 28657871
- [Background] Sampaio-Junior B, Tortella G, Borrione L, Moffa AH, Machado-Vieira R, Cretaz E, Fernandes da Silva A, Fraguas R, Aparicio LV, Klein I, Lafer B, Goerigk S, Bensenor IM, Lotufo PA, Gattaz WF, Brunoni AR. Efficacy and Safety of Transcranial Direct Current Stimulation as an Add-on Treatment for Bipolar Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Feb 1;75(2):158-166. doi: 10.1001/jamapsychiatry.2017.4040. PMID 29282470
- [Background] Tavares DF, Suen P, Rodrigues Dos Santos CG, Moreno DH, Lane Valiengo LDC, Klein I, Borrione L, Marques Forte P, Brunoni AR, Alberto Moreno R. Treatment of mixed depression with theta-burst stimulation (TBS): results from a double-blind, randomized, sham-controlled clinical trial. Neuropsychopharmacology. 2021 Dec;46(13):2257-2265. doi: 10.1038/s41386-021-01080-9. Epub 2021 Jun 30. PMID 34193961
- [Background] Silva RMFD, Brunoni AR, Goerigk S, Batistuzzo MC, Costa DLDC, Diniz JB, Padberg F, D'Urso G, Miguel EC, Shavitt RG. Efficacy and safety of transcranial direct current stimulation as an add-on treatment for obsessive-compulsive disorder: a randomized, sham-controlled trial. Neuropsychopharmacology. 2021 Apr;46(5):1028-1034. doi: 10.1038/s41386-020-00928-w. Epub 2021 Jan 15. PMID 33452434
- [Background] Valiengo LDCL, Goerigk S, Gordon PC, Padberg F, Serpa MH, Koebe S, Santos LAD, Lovera RAM, Carvalho JB, van de Bilt M, Lacerda ALT, Elkis H, Gattaz WF, Brunoni AR. Efficacy and Safety of Transcranial Direct Current Stimulation for Treating Negative Symptoms in Schizophrenia: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Feb 1;77(2):121-129. doi: 10.1001/jamapsychiatry.2019.3199. PMID 31617873
- [Background] Beam W, Borckardt JJ, Reeves ST, George MS. An efficient and accurate new method for locating the F3 position for prefrontal TMS applications. Brain Stimul. 2009 Jan;2(1):50-4. doi: 10.1016/j.brs.2008.09.006. PMID 20539835
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Vilela JA, Crippa JA, Del-Ben CM, Loureiro SR. Reliability and validity of a Portuguese version of the Young Mania Rating Scale. Braz J Med Biol Res. 2005 Sep;38(9):1429-39. doi: 10.1590/s0100-879x2005000900019. Epub 2005 Aug 26. PMID 16138228
- [Background] Li CT, Chen MH, Juan CH, Huang HH, Chen LF, Hsieh JC, Tu PC, Bai YM, Tsai SJ, Lee YC, Su TP. Efficacy of prefrontal theta-burst stimulation in refractory depression: a randomized sham-controlled study. Brain. 2014 Jul;137(Pt 7):2088-98. doi: 10.1093/brain/awu109. Epub 2014 May 10. PMID 24817188
- [Derived] Ramos MRF, Goerigk S, Aparecida da Silva V, Cavendish BA, Pinto BS, Papa CHG, Resende JV, Klein I, Carneiro AM, de Sousa JP, Vidal KSM, Valiengo LDCL, Razza LB, Aparicio LM, Martins L, Borrione L, Batista M, Moran NK, Dos Santos LA, Benatti R, Pelosof R, Padberg F, Brunoni AR. Accelerated Theta-Burst Stimulation for Treatment-Resistant Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2025 May 1;82(5):442-450. doi: 10.1001/jamapsychiatry.2025.0013. PMID 40042840
- See also: Organization World Health, Others. Depression and other common mental disorders: global health estimates. World Health Organization; 2017. — https://apps.who.int/iris/bitstream/handle/10665/254610/WHO-MSD-MER-2017.2-eng.pdf